CLINICAL TRIAL: NCT04987814
Title: HD-sEMG Markers of Sarcopenia
Brief Title: High-definition Surface Electromyography Markers for the Diagnosis of Sarcopenia
Acronym: CHRONOS-SARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP201339
Record Dates: First submitted 2021-04-29; First posted 2021-08-03 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
Keywords: High definition surface electromyography; Sarcopenia; Muscle; Biphotonic X-ray absorptiometry; Dual x-ray absorptiometry (DEXA)
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly patients suspected of sarcopenia (Experimental)
  Interventions: Other: HD-sEMG; Other: - Quadriceps muscle ultrasound; Other: IPAQ Physical Activity Questionnaire.

INTERVENTIONS:
Other: HD-sEMG — high definition surface electromyography, allowing the recording of muscle activation signals sensitive to the intensity of the contraction and indirectly to the muscle strength as well as to the muscular fatigability, but also capable of measuring the modifications of the recruitment modalities of the motor units. This recording will be made on the rectus femoris during knee extension, either in the lying position or during chair lifts, depending on the patient's functional state.
Other: - Quadriceps muscle ultrasound — Muscle Ultrasound with Philips Lumify Wireless Handheld Ultrasound for Android - Model - L12-4 linear probe, allowing performance at the patient's bed.
Other: IPAQ Physical Activity Questionnaire. — physical activity assessment questionnaire/adapted version for seniors

SUMMARY:
Sarcopenia is a progressive and generalised skeletal muscle disorder involving the accelerated loss of muscle mass and function that is associated with increased adverse outcomes including falls, functional decline, frailty, and mortality.

In this pilot project, the investigators want to explore the potential of the high-definition surface electromyography technology (HD-sEMG) for the diagnosis of sarcopenia.

This is a monocentric, descriptive, cross-sectional, parallel group study to develop a new diagnostic method.

It is planned to include 50 people aged 75 years and over hospitalized in the acute geriatric ward and suspected of sarcopenia (Score ≥4 on the SARC-F screening questionnaire).

The inclusion duration will be 36 months and adding a 1-month patient follow-up as part of routine care, the total study duration will be 37 months.

Patients will have their body composition (muscle mass, fat mass, and bone mass) using dual X-ray absorptiometry (DEXA). Muscular strength will be assessed by handgrip strength. Physical performance will be assessed. Additional data will be collected from their medical records.

DETAILED DESCRIPTION:
The aging of the population is a major public health problem with its multifactorial impact on quality of life and maintenance of autonomy. Unfortunately, one consequence of aging is sarcopenia, which affects the intrinsic and functional properties of muscle. It is a risk factor for loss of autonomy, falls, frailty and is associated with increased mortality.

Sarcopenia is defined as a progressive loss of muscle mass, strength and physical performance. Classically, sarcopenia is assessed by imaging techniques (MRI, DEXA) or bioelectrical impedancemetry for aspects related to the assessment of muscle mass loss. MRI or DEXA are not widely available and/or access is limited.

For functional aspects, grip strength measurements are often used. Currently sarcopenia cannot be diagnosed and evaluated by a single examination, including both the morphological (muscle mass) and functional aspects. Furthermore, several biological markers are associated with muscle mass, strength, and function, but these biomarkers are not specific to skeletal muscle and are weakly associated with clinical goals.

Finally, despite the important interest in assessing the qualitative/functional and quantitative aspect of skeletal muscle in neuromuscular impairment, there is currently no tool that routinely assesses these aspects.

In this context, developing new approaches for non-invasive assessment of sarcopenia, is a major issue. In this pilot project, the investigators aim to develop a medical device derived from high-definition surface electromyography (HD-sEMG) technology, non-invasive and portable, for the diagnosis of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 years and over
* Score ≥4 on the SARC-F screening questionnaire
* Enrolled in a social security plan (no AME)
* Informed and consenting patient

Exclusion Criteria:

* BMI ≥30 kg/m2
* Untreated/unbalanced endocrinological pathology
* Myopathy
* Inflammatory or autoimmune pathology
* Severe psychiatric pathology or severe cognitive disorders that do not allow the performance of examinations
* Patients who are dependent for all acts of daily life
* Patients with a very short life expectancy
* Recent fracture or trauma of the lower limbs preventing dynamic measurement of HD-sEMG recording
* Bilateral hip prosthesis
* Skin problem that may interfere with the recording of surface EMG activity
* Patient under guardianship / curatorship

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Electromyographic signals of the rectus femoris collected by the HD-sEMG technique | day1-day7
  These signals will be confronted by the diagnosis of sarcopenia defined by the joint presence of the 2 clinical criteria of the European Working Group on Sarcopenia in Older People 2 (EWGSOP2).

SECONDARY OUTCOMES:
Number of participants with falls. Definition of " fallers " : at least 1 fall in the last 12 months | day1- day7
  Information will be collected in the medical record.
Skeletal muscle mass index (SMMI in kg/m2, skeletal muscle mass/height2) collected by DEXA | day1-day7
Grip strength by dynamometer (kg) | day1-day7
SPPB score (SHORT PHYSICAL PERFORMANCE BATTERY score) | day1-day7
  Short Physical Performance Battery (SPPB): score range 0-12, higher score means a better outcome
HD-sEMG muscle data, measured during lower limb quadriceps extension by High Definition Surface Electromyography HD-sEMG | 1 month post inclusion
  HD-sEMG parameters will be collected by HD-sEMG technique with TMSi's Mobita equipment, CE marked (European compliance). They will be collected by electrical measurements from a grid of electrodes (32 channels) placed on the muscle surface. The results of the measurement will be represented by a muscle activation mapping.
Rate of Mortality at 1 month | 1 month post inclusion
  Rate of participants who deceased at 1 month. Mortality will be measured with vital status at 1 month.
Muscle and subcutaneous fat thicknesses of the quadriceps in mm | day1-day7
  Muscle and subcutaneous fat thickness of the quadriceps in mm evaluated by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoka KINUGAWA, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - Service de gériatrie aigue polyvalente (GAP), Ivry-sur-Seine
  - Service de soins de suite et de réadaptation Gériatrique 1, Ivry-sur-Seine
  - Service de soins de suite et de réadaptation gériatrique 2, Ivry-sur-Seine
  - Unité d'Explorations fonctionnelles du sujet âgé, Hôpital Charles Foix, Ivry-sur-Seine
  - Service de soins de suite et de réadaptation -Plaies et cicatrisation, Paris
  - Service de soins de suite et de réadaptation Gériatrique Hôpital Rothschild, Paris

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal